CLINICAL TRIAL: NCT00039104
Title: A Phase II, Open-Label, Randomized Trial of Zoledronic Acid (Zometa™) and BMS-275291 (NSC#713763) in Patients With Hormone Refractory Prostate Cancer
Brief Title: Zoledronate and BMS-275291 in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02799; MC0151; N01CM17104 (NIH)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-((2S)-2-mercapto-1-oxo-4-(3,4,4- trimethyl-2,5-dioxo-1-imidazolidinyl)butyl)-L-leucyl-N,3- dimethyl-L-Valinamide; Zoledronic Acid

ARMS (2):
- Arm I (rebimastat, zoledronic acid) (Experimental): Patients receive zoledronate IV over at least 15 minutes on day 1 and oral BMS-275291 daily on days 1-28.
  Interventions: Drug: rebimastat; Drug: zoledronic acid; Other: laboratory biomarker analysis
- Arm II (zoledronic acid) (Experimental): Patients receive zoledronate as in Arm I.
  Interventions: Drug: zoledronic acid; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: rebimastat — Given PO
  Other Names: BMS-275291; D2163
  Arms: Arm I (rebimastat, zoledronic acid)
Drug: zoledronic acid — Given IV
  Other Names: CGP 42446; CGP42446A; NDC-zoledronate; zoledronate; Zometa
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining zoledronate with BMS-275291 in treating patients who have prostate cancer that has not responded to previous hormone therapy. Zoledronate may prevent bone loss and stop the growth of tumor cells in bone. BMS-275291 may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth. Combining zoledronate with BMS-275291 may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the confirmed response rate of hormone refractory prostate cancer patients treated with Zometa with BMS-275291.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile associated with this treatment in this patient population.

II. To evaluate the overall and progression-free survival associated with this treatment regimen.

III. To explore changes markers for bone turnover, fPYR, fDPYR, and serum samples for cross-linked N-telopeptides from baseline.

IV. To assess changes in bone tumor metabolism after treatment using PET scans. V. To assess changes in MMP-1, MMP-9, VEGF and bFGF from baseline after treatment.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to prior chemotherapy (yes vs no) and participating center.

ARM I: Patients receive zoledronate IV over at least 15 minutes on day 1 and oral BMS-275291 daily on days 1-28.

ARM II (CLOSED TO ACCRUAL AS OF 10/10/2003): Patients receive zoledronate as in Arm I.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed (adeno)carcinoma of the prostate refractory to hormone therapy
* Metastatic bone disease, as documented by bone scan and confirmed by x-rays, CT scan or MRI scan

  * Note: Patients may also have measurable disease in the lymph nodes (retroperitoneal, pelvic or inguinal only), prostate and /or prostatic bed; measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm =< 21 days prior to registration
* PSA progression defined as two consecutive increases in PSA value over the previous reference value; the first increase of PSA should occur no earlier than one (1) week after the reference measurement; all patients need to demonstrate continued PSA elevation with an increasing PSA four weeks after the required cessation of their antiandrogen treatment; the required cessation period is 4 weeks for flutamide, nilutamide, and Megace-based treatment, and 8 weeks for bicalutamide-based treatment
* One of the following:

  * Continuing primary androgen suppression (LHRH agonist)
  * Orchiectomy
* WBC >= 2000/mm^3
* Absolute neutrophil count (ANC) >= 1500/mm^3
* PLT >= 100,000/mm^3
* Hgb >= 9.0 g/dL
* Total bilirubin =< institutional upper normal limits (UNL)
* AST =< 1.5 x UNL
* Serum creatinine =< 1.5 x UNL
* PSA >= 5 ng/mL
* Serum testosterone < 50 ng/dL =< 3 months prior to registration
* Estimated life expectancy of >= 6 months
* ECOG Performance Status (PS) 0, 1, or 2
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent
* If sexually active, willing to use an accepted and effective method of contraception consistently for the duration of study participation

Exclusion Criteria:

* Any of the following:

  * > 2 prior chemotherapy regimen
  * > 2 non-hormonal treatments for metastatic disease (including biologics, gene therapy, angiogenesis inhibitors, etc., but excluding external radiotherapy)
  * Prior therapy with a matrix metalloproteinase inhibitor (MMPI)
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Radiation therapy =< 4 weeks prior to study entry
  * Concomitant hormonal treatment (except LHRH)
  * Prior use of systemic radiopharmaceuticals such as samarium and strontium
  * PC-Spes =< 4 weeks prior to study entry
  * Failure to fully recover from adverse effects of prior therapies regardless of interval since last treatment
  * Other concurrent chemotherapy, immunotherapy, or radiotherapy directed at the cancer
  * Other therapy or supportive care that is considered investigational
* Known CNS metastases
* Known visceral metastases (pulmonary, liver, kidney, splenic lesions); patients with retroperitoneal, pelvic or inguinal lymph node metastases and/or disease in the prostate (or prostatic bed) will not be excluded
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancer from which the patient has been disease free for >= 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-04; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Confirmed response (PSA decline of greater than 50% confirmed at least four weeks apart) | Up to 2 years

SECONDARY OUTCOMES:
Overall survival time | From registration to death due to any cause, assessed for up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | From registration to documentation of disease progression, assessed up to 2 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of PSA response or duration of PSA control | Up to 2 years
  The distribution of this response duration will be estimated using the method of Kaplan-Meier.
Incidence of toxicity as per NCI CTCAE version 2.0 | Up to 2 years
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States